CLINICAL TRIAL: NCT04218799
Title: Human Microbiome and Healthcare Associated Infections - Nursing Home Dwelling Older Veterans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary-Claire Roghmann, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HP-00058923
Record Dates: First submitted 2019-12-20; First posted 2020-01-06 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Human Microbiome
Keywords: intranasal mupirocin; topical chlorhexidine
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intranasal Mupirocin and Topical Chlorhexidine (Experimental)
  Interventions: Drug: Intranasal Mupirocin and Topical Chlorhexidine

INTERVENTIONS:
Drug: Intranasal Mupirocin and Topical Chlorhexidine — Antimicrobial antiseptic skin cleanser (4% chlorhexidine) for daily use on Day 1, 3 and 5 of Week 8 of the study. BACTROBAN NASAL ointment (mupirocin calcium ointment, 2%) for use intranasally twice-daily on Day 1, 2, 3, 4 and 5 of Week 8 of the study.

SUMMARY:
The purpose of the research is to find out the effect of commonly used topical antibiotics on the bacteria that live in the nose, throat and on the skin of older adults. In addition, the investigators want to determine if these topical antibiotics affect how bacteria are spread in Community Living Centers of the VA Maryland Health Care System.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older.
* Living in a participating nursing home for at least 80% of the past 3 months-
* Willing to provide anterior nares, posterior pharynx, skin and throat specimens over the study period.
* Willing to use intranasal mupirocin and topical chlorhexidine over a five day period.
* Provide signed and dated informed consent from subject or LAR.

Exclusion Criteria:

* Recent history of MRSA colonization
* Use of mupirocin nasal ointment in past 3 months
* Use of topical chlorhexidine in past 3 months
* History of an allergic reaction to chlorhexidine or mupirocin

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2015-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Claire Roghmann, MD, MS, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - Loch Raven VA Community Living Center, Baltimore, Maryland
  - Perry Point VA Community Living Center, Perry Point, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants were S. aureus negative in the nose at enrollment and were withdrawn from the study as the use of mupirocin was not clinically indicated. 1 participant was discharged from the nursing home prior to receiving mupirocin.
Period: Overall Study
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in the Abundance of Staphylococcus Aureus in the Nose After Decolonization
Description: Change in the abundance of Staphylococcus aureus in the nose from immediately before mupirocin administration to 8 weeks after mupirocin administration.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: fg/uL
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 7
fg/uL | -4174 (11003)

2. Primary Outcome: Change in the Abundance of Staphylococcus Aureus in the Throat After Decolonization
Description: Change in the abundance of Staphylococcus aureus in the throat from immediately before mupirocin administration to 8 weeks after mupirocin administration.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: fg/uL
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 7
fg/uL | -3395 (8954)

3. Primary Outcome: Change in the Abundance of Gram Negative Bacteria on the Subclavian Skin After Decolonization
Description: Quantitative PCR using 16s rRNA is used to quantify the total bacterial load of Gram negative bacteria on the subclavian skin before and after decolonization.
Time Frame: 12 months
Population: Subclavian skin samples deteriorated prior to sample analysis and cannot be used.
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 0

4. Primary Outcome: Change in the Abundance of Gram Negative Bacteria on the Femoral Skin After Decolonization
Description: Quantitative PCR using 16s rRNA is used to quantify the total bacterial load of Gram negative bacteria on the femoral skin before and after decolonization.
Time Frame: 12 months
Population: Femoral skin samples deteriorated prior to sample analysis and cannot be used.
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Intranasal Mupirocin and Topical Chlorhexidine
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes